

# Statistical Analysis Plan (SAP) BCG-DENMARK-ELDERLY

## Part A:

Using BCG vaccine to enhance non-specific protection of senior citizens during the COVID-19 pandemic. A randomized clinical trial (BCG-DENMARK-SENIOR).

## Part B:

Using BCG vaccine to strengthen the immune system in the elderly and improve the response to influenza vaccine. A randomized clinical trial (BCG-DENMARK-INFLUENZA).







## **TABLE OF CONTENTS**

| PART A | Page 3-20 |
|-------------------------------------------|------------|
| 1.0 Administrative information | Page 3 |
| 2.0 Introduction | Page 4 |
| 3.0 Study methods | Page 4 |
| 4.0 Statistical principles | Page 5 |
| 5.0 Study population | Page 6 |
| 6.0 Description of outcomes and variables | Page 6 |
| 7.0 Analysis | Page 8 |
| 8.0 Supplementary information | Page 11 |
| PART B | Page 21-40 |
| 1.0 Administrative information | Page 21 |
| 2.0 Introduction | Page 22 |
| 3.0 Study methods | Page 23 |
| 4.0 Statistical principles | Page 24 |
| 5.0 Study population | Page 24 |
| 6.0 Description of outcomes and variables | Page 25 |
| 7.0 Analysis | Page 28 |
| 8.0 Supplementary information | Page 29 |
| 9.0 References | Page 41-42 |





# 1.0 ADMINISTRATIVE INFORMATION, Part A

| Title | Using BCG vaccine to enhance non-specific protection of senior citizens during the COVID-19 pandemic. A randomized clinical trial (BCG- |
|---|---|
| | DENMARK-SENIOR). |
| Trial registration | EudraCT number 2020-003904-15 |
| SAP version and date | 2.0, 08-06-2023 |
| Protocol version and date | 4.3, 31-01-2022 |
| SAP contributors | Anne Marie Rosendahl Madsen (PI) |
| | Christine Stabell Benn (Sponsor) |
| | Lise Gehrt (Data analyst) |
| | Ola Løvsletten (Statistician) |
| Sponsor | Christine Stabell Benn |
| | University of Southern Denmark, Department |
| | of Clinical Research and Bandim Health Projec |
| Primary investigator | Anne Marie Rosendahl Madsen |
| | University of Southern Denmark, Department |
| | of Clinical Research and Bandim Health Projec |
| Trial statistician | Ola Løvsletten |
| | The Arctic University of Norway, Tromsø |
| | Department of Community medicine |
| SAP revision history | Revision 08-06-2023: |
| | Updated section 6.0 and 7.0: |
| | 1. The composite outcome will include all |
| | infectious disease hospital contacts. |
| | 2. Data does not support analysis of COVID-19 |
| | severity, this outcome has been removed. |
| | 3. New secondary outcome has been added: |
| | All-cause hospitalization. |





## 2.0 INTRODUCTION

## Background

Worldwide, the population of persons > 60 years of age is growing because of advances in average life expectancy, especially in high income countries<sup>[1]</sup>. Due to age related decline in immune function, so called immunosenescence, the elderly are at higher risk of infectious diseases<sup>[2]</sup>. Severe infections are more common in the elderly, and they are more likely to be hospitalized due to complications related to infectious diseases. During the COVID-19 pandemic, it has become clear that elderly people are particularly susceptible to severe COVID-19. Strategies to strengthen senior citizens' immune system are urgently warranted.

The Bacille Calmette Guérin (BCG) vaccine was developed for tuberculosis prevention, but there is increasing evidence that it also has beneficial heterologous "non-specific" effects on the immune system<sup>[3–5]</sup>. Prior studies have shown that BCG vaccination strengthens the innate immune system resulting in increased activity against non-related infections<sup>[6–8]</sup>. BCG vaccination may strengthen the immune system of senior citizens and may (partially) protect against getting infected and/or experiencing severe morbidity due to infections in general and SARS-CoV-2 in particular<sup>[9,10]</sup>.

We hypothesize that BCG vaccination can reduce the risk of COVID-19 and other infections among senior citizens during the COVID-19 pandemic<sup>[11]</sup>. A randomized controlled trial provides the highest validity for this research question.

## **Objectives and hypothesis**

Primary objective: To reduce senior citizens' risk of acute infection during the COVID-19 pandemic.

Secondary objectives: To reduce senior citizens' risk of SARS-CoV-2 infection during the COVID-19 pandemic and to reduce self-reported respiratory illness in general during the COVID-19 pandemic.

The hypothesis is that BCG vaccination of seniors will reduce the risk of acute infection by 25% over a period of 12 months.

#### **3.0 STUDY METHODS**

#### **Trial design**





A single-blinded, placebo controlled randomized clinical trial. Participants are randomized 1:1 to BCG or placebo and will be followed for 12 months post-randomization with respect to illness, medical contacts, use of antibiotics, hospitalization, and death. The follow-up takes place both through self-reporting and through the Danish National Registers. The participants will receive an electronic questionnaire biweekly with questions about illness, medical contacts, other vaccinations, and side effects.

People ≥ 65 years of age are eligible for participation.

#### Randomization

Randomization takes place at baseline after informed consent is given. The randomization is done in varying blocks of 6-8, stratified by sex and age group (65-74; 75+) using REDCap electronic data capture tools hosted at the Region of Southern Denmark<sup>[12,13]</sup>.

#### Sample size

With an expected incidence of "acute infection" of 20% we will be able to show a 25% reduction in the risk of acute infection in the intervention group compared to the placebo group by including a total of 1890 individuals: 945 individuals in each group. Since the primary outcome data to a large extent are obtained via national registers, we anticipate limited loss of power due to loss to follow-up. We therefore aimed to enroll 1900 participants.

Due to the pandemic and varying infectious disease precautions, recruitment took longer than anticipated, and we ended up recruiting a total of 1706 participants (90% of the anticipated sample size) between September 2020 and December 2021.

## Timing of final analyses and outcome assessments

All outcomes are analyzed after end of trial.

#### 4.0 STATISTICAL PRINCIPLES

#### Levels of confidence and p-values

A double-sided p-value of < 0.05 will be considered statistically significant. 95% confidence intervals will be provided.

#### **Protocol violations**





Protocol deviations and exclusions will be reported for each treatment arm.

#### **5.0 STUDY POPULATION**

#### Screening data

Around 35,000 elderly > 65 years live in Odense at the time of recruitment. The study is based on voluntary participation open to all eligible persons on their own initiative. Interested persons are screened for participation after they have received oral and written information and declared their continued interest for participation. We keep a list of persons screened for participation and reasons for not being included/being excluded.

#### Recruitment

Recruitment, enrolment, and follow-up with collection of biological material is conducted at activity houses for senior citizens run by the Municipality of Odense. The project is presented at special arrangements at these houses and advertised in local media and via posters in relevant public places.

#### Exclusion/loss to follow-up

Participants who are excluded after randomization or lost to follow up are not replaced.

Participants are under follow-up for 12 months post-randomization or until they withdraw their consent, migrate to another country, or die.

#### Baseline characteristics, study population

Continuous baseline characteristics will be reported as mean with standard deviation or median with inter-quartile range, as appropriate. Categorical baseline characteristics will be reported as count and percentage. No statistical testing for baseline characteristics will be performed.

#### **6.0 DESCRIPTION OF OUTCOMES AND VARIABLES**

## **Primary outcome**

The primary outcome is a composite outcome: acute infection identified either by a doctor, by antibiotics use, by hospitalization, or by death due to infection. All subcomponents will also be presented separately.





Information on hospitalizations, deaths, and antibiotics use is retrieved from national health registers: The Danish National Patient Register, The Central Person Register, and The National Prescription Register. All hospital contacts due to acute infection will be included, regardless of duration of the contact. An acute infection event identified by a doctor is defined as newly onset infectious illness that has prompted the participant to seek medical attention from general practitioner (GP) or on-call doctor and is based on self-reporting. Participants are asked in the questionnaires, if they have needed to see their GP or an on-call doctor due to newly onset illness during the past 14 days (yes/no). Thus, participants can only have one such event per survey period (14 days). For all outcomes, a honeymoon period of 14 days will be used to define new events.

#### **Secondary outcomes**

Secondary outcomes are verified SARS-CoV-2 infection (first event), self-reported respiratory infection, and all-cause hospitalization (first event). Information on positive test results will be retrieved from the Danish Health Data Authority (Sundhedsdatastyrelsen) and information on self-reported respiratory infections will come from the follow-up questionnaires.

Verified SARS-CoV-2 infection is defined as having a positive SARS-CoV-2 PCR (Polymerase Chain Reaction), rapid antigen test, or converting from negative to positive antibody test (IgG positive) without having been vaccinated.

Self-reported illness is defined as a respiratory infection if the participants report having had a respiratory infection such as common cold, influenza, pneumonia or similar term, or they report having had one or more of the following symptoms: cough, sore throat, runny nose/nasal congestion (common cold symptoms), loss of smell or taste sense, or dyspnea with or without general symptoms such as fever, chills, muscle ache, headache, and fatigue (dyspnea only if in combination with fever).

All-case hospitalization (first event) will include all hospital contacts with duration of 24 h or more, to ensure we only include hospital admissions and not visits to outpatient clinics.





## **Variables**

| Variable | Definition | Туре | Scale |
|---|---|---|---|
| Primary outcome: | | | |
| Acute infection | Death, hospitalization, antibiotic | Categorical, binary | 0,1 |
| | treatment, or visit to GP due to | | |
| | newly onset infectious disease. | | |
| | Composite outcome. | | |
| Death due to | Death due to infectious disease. | Categorical, binary | 0,1 |
| infection | | | |
| Hospitalization for | Hospital contact due to infectious | Categorical, binary | 0,1 |
| infection | disease. | | |
| Antibiotic | Antibiotic treatment during Categorical, bir | | 0,1 |
| treatment | follow-up. | | |
| Doctor diagnosed | Infection identified by GP or on- | Categorical, binary | 0,1 |
| infection | call doctor. | | |
| Secondary outcomes: | | | |
| Self-reported | Reported respiratory symptoms | Categorical, binary | 0,1 |
| respiratory infection | or disease compatible with | | |
| | respiratory infection. | | |
| Verified CoV <sup>1</sup> | Positive SARS-CoV-2 test. | Categorical, binary | 0,1 |
| infection (first event) | | | |
| All-cause | Admission to hospital > 24 hours | Categorical. binary | 0, 1 |
| hospitalization | (first event). | | |

<sup>&</sup>lt;sup>1</sup> SARS-CoV-2 infection.

## 7.0 ANALYSIS

## Methods

All analyses will be performed from the intention-to-treat principle, for all participants studied together and stratified by sex and age group.

Several couples participated in this study. To consider shared vulnerability, we will cluster on couples (non-stratified analysis).

## **Primary outcome:**

Acute infection will be analyzed as a recurrent time-to-event using an Andersen-Gill Cox proportional hazards regression model with time since inclusion as underlying time scale. The proportional hazards assumption will be tested using Schoenfeld residuals. The analysis





will be done for the composite outcome and for all the subcomponents separately presenting hazard ratio with 95% confidence intervals for each. Absolute risk reductions will be calculated using Cox regression.

## **Secondary outcomes:**

The secondary endpoint self-reported respiratory infection will be analyzed the same way as the primary endpoint. As participants are only able to report one infectious episode during a follow-up questionnaire, the event will be assigned to the first day within the questionnaire period, and the following 14 days of follow-up excluded for analyses as it represents risk free time.

The secondary outcomes verified SARS-CoV-2 infection and all-cause hospitalization will be analyzed in a standard Cox proportional hazards model, but otherwise as described above.

## **Supplementary analyses**

We will conduct preplanned supplementary analyses to assess possible effect modification by other vaccines given during follow-up, previous BCG vaccination, and COVID-19 vaccination before inclusion. These will be done using the same methods as described above for the primary (composite) outcome and for all secondary outcomes.

1. Before and after receipt of subsequent vaccines, and adjusted by type of subsequent vaccine, to assess possible interaction between BCG and other vaccines. Vaccination status will be categorized as 1) No other vaccines, 2) COVID 19 vaccine, 3) Influenza vaccine, or 4) COVID 19 and influenza vaccine.

Vaccination status will be included as a time varying covariate changing on the date of vaccination with subsequent vaccines received during follow-up. Some participants received a pneumococcal vaccine (23-valent polysaccharide vaccine) together with their influenza vaccine as was recommended by the Danish Board of Health in 2020. We will therefore include influenza vaccines with or without concurrent pneumococcal vaccination (given on the same day). Participants will be censored upon receipt of any other vaccines than the above mentioned.

2. By previous BCG vaccination (Yes/no, self-reported and assessed by BCG scar) to assess the effect of revaccination vs. first vaccination with BCG.





3. By COVID-19 vaccination status at inclusion (Received COVID 19 vaccines yes/no).

## **Exploratory analysis**

Participants were enrolled during different stages of the COVID-19 pandemic. We will therefore conduct a subgroup analysis of all outcomes comparing participants included in the same phase of the pandemic. We will compare outcomes for participants included in the following periods:

- September 2020 to January 2021 (N=1239); before the COVID-19 vaccines were widely distributed to the target population. A period characterized by increasing infection control measurements and concluding in lockdown.
- 2. April to December 2021 (N=438); Participants are now being vaccinated with the new coronavirus vaccines; most have had the two or three doses before enrollment. A period characterized by varying COVID-19 activity; a minimum of restrictions on society despite periodically high transmission rates (Omicron variant in the fall).

## Missing data

Participants are under follow-up for the primary outcome irrespective of missing questionnaires as this is mostly based on register data.

For the outcomes solely based on self-reported information (self-reported respiratory infections and severity of COVID-19) participants are only under follow-up during the periods where they have completed follow-up questionnaires.

#### **Adverse events**

Adverse events will be described in terms of incidence in the groups and more thoroughly presented in a table as part of supplementary material (Table 4). Serious adverse events (SAE) will be classified as related to study drugs (possible/probable/definite) or unrelated to study drugs (unlikely/doubtful). If related, they are classified as expected/unexpected (SAR/SUSAR).

#### 8.0 SUPPLEMENTARY INFORMATION

## Figures and tables

Figure 1: Flow chart, inclusion.







Table 1: Baseline characteristics.

Table 2: Results primary and secondary outcomes.

Table 3: Supplementary analyses (sex, age group, other vaccines, previous BCG, COVID-19

vaccination status at inclusion).

Table 4: Adverse events and serious adverse events.

Table 5: Short description of serious adverse events.





Figure 1: Flow chart, inclusion

## **CONSORT 2010 Flow Diagram**





# **Table 1 Baseline characteristics**

| | BCG | Placebo |
|-------------------------------------------|-----|---------|
| Age, median (IQR) | | |
| Sex female (%) | | |
| Living alone (%) | | |
| Spouse included in study (%) | | |
| Active smoker (%) | | |
| Previous smoker (%) | | |
| Alcohol consumption, units per week, mean | | |
| (SD) | | |
| BMI, median (IQR) | | |
| Chronic diseases | | |
| Cardiovascular (%) | | |
| Diabetes (%) | | |
| Lung (%) | | |
| Other (%) | | |
| Level of education | | |
| Low (%) | | |
| Medium (%) | | |
| High (%) | | |
| Previously BCG vaccinated (%) | | |
| Scar from BCG vaccination observed (%) | | |
| COVID-19 vaccinated, yes (%) <sup>1</sup> | | |
| One dose | | |
| Two doses | | |
| Three doses | | |

<sup>&</sup>lt;sup>1</sup>COVID-19 vaccinated before enrollment.





# Table 2 Results primary and secondary outcomes

| Outcome | Numb | er (%) | Hazard ratio | Absolute risk |
|---|---|---|---|---|
| | BCG | Placebo | (95% CI) | reduction |
| | N=xxx | N=xxx | | (95% CI) |
| Primary outcome | | | | |
| Acute infection | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Death | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Hospitalization | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Antibiotics | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Doctor | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Secondary outcomes | | | | |
| - | | | | |
| Self-reported | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| respiratory | | | | |
| infection | | | | |
| Verified COVID-19 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| All-cause<br>hospitalization | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |



Table 3 Supplementary analyses to explore possible effect modification by sex, age group, other vaccines, previous BCG, and COVID-19 vaccination status at inclusion.

| | Nun | nber (%) | Hazard ratio | Absolute risk |
|---|---|---|---|---|
| | BCG | Placebo | (95% CI) | reduction |
| | N=xxx | N=xxx | | (95% CI) |
| Acute infection – also wl | nere num | bers permit s | ubdivided on each o | of the outcomes |
| included in the composit | e outcom | e. | | |
| Females | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Males | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Age < 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Age ≥ 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Other vaccines received after randomization: Effect of | | | | |
| intervention before<br>other vaccines<br>Effect of | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| intervention after other vaccines | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Effect after other vaccines, by type of vaccine received: | | | | |
| COVID vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| Influenza vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| Both vaccines | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| Has BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| No BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| CoV vaccinated before enrollment: | | | | |
| Yes | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| No | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| Included period 1 <sup>2</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Included period 2 <sup>3</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |



| Self-reported respiratory | / infection | | | |
|---|---|---|---|---|
| Females | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Males | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Age < 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Age ≥ 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Other vaccines received | | | | |
| after randomization: | | , , | , , | |
| Effect of | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| intervention before | | | | |
| other vaccines | | | | |
| Effect of | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| intervention after | | | | |
| other vaccines | | | | |
| Effect after other | | | | |
| vaccines, by type of | | | | |
| vaccine received: | | | | |
| COVID vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Influenza vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Both vaccines | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Has BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| No BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| CoV vaccinated before | | | | |
| enrollment: | | | | |
| Yes | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| No | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| Included period 1 <sup>2</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Included period 2 <sup>3</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Verified COVID-19 | | | | |
| Females | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Males | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Age < 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Age ≥ 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |





| 011 | | | | |
|---|---|---|---|---|
| Other vaccines received | | | | |
| after randomization: | | | | |
| Effect of | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| intervention before | | | | |
| other vaccines | | | | |
| Effect of | | | | |
| intervention after | xx (x.x) | xx (x.x) | x.xx (x.xx-x.xx) | x.x% (x.x%-x.x%) |
| other vaccines | , , | ` ' | , | , |
| Effect after other | | | | |
| vaccines, by type of | | | | |
| vaccine received: | | | | |
| | | () | | 0/ /0/0/\ |
| COVID vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Influenza vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Both vaccines | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Has BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| No BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| CoV vaccinated before | | | | |
| enrollment: | | | | |
| Yes | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| No | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Included period 1 <sup>2</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Included period 2 <sup>3</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| All-cause hospitalization | | | | |
| Females | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| T CITICIO | 70. (70.7.) | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | Allow (Allow Allow) | Allaye (Allaye Allaye) |
| Males | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Age < 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Age ≥ 75 | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Other vaccines received | | | | |
| after randomization: | | | | |
| Effect of | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| intervention before | | (*****) | | (1111/07/111/07 |
| other vaccines | | | | |
| Effect of intervention | | | | 0/ /0/ |
| after other vaccines | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |





## SAP BCG-DENMARK-ELDERLY, version 2.0, 08-06-2023

| Effect after other | | | | |
|---|---|---|---|---|
| vaccines, by type of | | | | |
| vaccine received: | | | | |
| COVID vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Influenza vaccine | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Both vaccines | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Has BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| No BCG scar <sup>1</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| CoV vaccinated before | | | | |
| enrollment: | | | | |
| Yes | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| No | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Included period 1 <sup>2</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%-x.x%) |
| Included period 2 <sup>3</sup> | xx (x.x) | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |

<sup>&</sup>lt;sup>1</sup>Scar from previous BCG vaccination at enrollment.



<sup>&</sup>lt;sup>2</sup> Period 1: September 2020 to January 2021 (N=1239); before the COVID-19 vaccines were widely distributed to the target population. A period characterized by increasing infection control measurements and concluding in lockdown.

<sup>&</sup>lt;sup>3</sup> Period 2: April to December 2021 (N=438); Participants are now being vaccinated with the new coronavirus vaccines; most have had the two or three doses before enrollment. A period characterized by varying COVID-19 activity; a minimum of restrictions on society despite periodically high transmission rates (Omicron variant in the fall).



# Table 4 Adverse Events (AE) and Serious Adverse Events (SAE)

| Any SAE Hospitalization for any reason Death due to any reason Adverse events (AE): Injection site reaction Minor abscess/wound | umber (%)<br>[M/F] | Number (%)<br>[M/F] |
|---|---|---|
| Hospitalization for any reason Death due to any reason Adverse events (AE): Injection site reaction | | |
| Death due to any reason Adverse events (AE): Injection site reaction | | |
| Adverse events (AE): Injection site reaction | | |
| Injection site reaction | | |
| Minor abscess/wound | | |
| Severe local reaction (abscess) | | |
| Fever | | |
| Fatigue | | |
| Headache | | |
| Lymphadenitis | | |
| Serious Adverse Events (SAE): | | |
| Blood or lymphatic disorder | | |
| Cardiac disorders | | |
| Endocrine disorders | | |
| Gastrointestinal disorders | | |
| Infection | | |
| Musculoskeletal and connective tissue disorders | | |
| Nervous system disorders | | |
| Respiratory disorders | | |





## SAP BCG-DENMARK-ELDERLY, version 2.0, 08-06-2023

| Urological and gynecological disorders |
|----------------------------------------|
| Unknown/other |
| Outcome SAE: |
| Life threatening |
| Required/prolonged hospitalization |
| Resulted in death |



# **Table 5 Short description of Serious Adverse Events (SAE)**

| No | Category | Outcome | Description | Group <sup>1</sup> | Sex | Week <sup>2</sup> | Before/after <sup>3</sup> |
|---|---|---|---|---|---|---|---|
| 1 | | | | | | | |
| 2 | | | | | | | |
| 3 | | | | | | | |
| 4 | | | | | | | |
| 5 | | | | | | | |
| 6 | | | | | | | |
| 7 | | | | | | | |
| 8 | | | | | | | |
| 9 | | | | | | | |
| 10 | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Randomisation group.

<sup>&</sup>lt;sup>2</sup>Weeks after inclusion.

<sup>&</sup>lt;sup>3</sup>Occurrence before or after other vaccines were administered to the participant.



# Statistical Analysis Plan (SAP)

| 1.0 ADMINISTRATIVE INFORMATION | ON, Part B |
|---|---|
| Title | Using BCG vaccine to strengthen the immune |
| | system in the elderly and improve the |
| | response to influenza vaccine. A randomized |
| | clinical trial (BCG-DENMARK-INFLUENZA). |
| Trial registration | EudraCT number 2019-002781-12 |
| SAP version and date | 1.0, 19-05-2023 |
| Protocol version and date | 5.6, 07-10-2021 |
| SAP contributors | Anne Marie Rosendahl Madsen (PI) |
| | Lise Gehrt (Data analyst) |
| | Ola Løvsletten (Statistician) |
| | Christine Stabell Benn (Sponsor) |
| Sponsor | Christine Stabell Benn |
| | University of Southern Denmark, Department |
| | of Clinical Research and Bandim Health Projec |
| Primary investigator | Anne Marie Rosendahl Madsen |
| | University of Southern Denmark, Department |
| | of Clinical Research and Bandim Health Projec |
| Trial statistician | Ola Løvsletten |
| | The Arctic University of Norway, Tromsø |
| | Department of Community medicine |
| SAP revision history | NA |
| Date of approval | 19-05-2023 (all authors). |



## 2.0 INTRODUCTION

## **Background**

Severe influenza virus infections are more common in the elderly and seasonal vaccination with inactivated influenza vaccine (IIV) is recommended to persons above 65 years of  $age^{[14]}$ . However, due to immunosenescence, the efficacy of vaccines decrease with increasing  $age^{[15,16]}$ .

The Bacille Calmette Guérin vaccine (BCG) was developed for tuberculosis prevention, but there is increasing evidence that it also has beneficial heterologous "non-specific" effects on the immune system<sup>[3,5,17]</sup>. Prior studies have shown that BCG vaccine strengthens the innate immune system resulting in increased activity against non-related infections<sup>[7,9,18]</sup>. A potentiating effect of BCG vaccine on the response to other vaccines has also been observed in previous studies<sup>[19–21]</sup>.

In the present project, we will explore BCG as a low-cost, low-risk intervention to increase the immune response to influenza vaccination and improve the general resistance towards infections in senior citizens.

#### **Objectives and hypothesis**

We will test the effects of BCG vaccination on the specific immune response to IIV and on the immune system and health in general in people  $\geq$  65 years, with the aim to:

- Improve their specific antibody response to influenza vaccination.
- Improve their general resistance towards infections.
- Study the effect of BCG on classical lymphocyte-dependent responses, and the induction of innate immune memory.

We will test the following hypotheses:

- a) BCG vaccine given two weeks prior to, together with, or two weeks after IIV is associated with a 30% increase in seroconversion to IIV and/or a significant increase in influenza antibody titers.
- b) The hypothesized potentiating effects of BCG is due to a combination of classical lymphocyte-dependent responses, and the induction of innate immune memory (trained





immunity) in myeloid cells.

#### **10.0 STUDY METHODS**

## **Trial design**

A single-blinded, placebo controlled, randomized clinical trial, with nested immunological studies. Participants are randomized 1:1:1:1 to four groups: BCG 14 days before, together with, or 14 days after IIV compared to placebo.

People ≥ 65 years of age who plan to accept the offer of seasonal influenza vaccination are eligible for participation.

Participants are vaccinated once at day 0 and twice at day 14 (one shot in each arm). All participants receive the standard seasonal IIV recommended by the Danish Board of Health. The participants will come back for a follow-up interview at day 42 and all are followed for six months post-randomization with electronic questionnaires about their health. These include information on symptoms and disease, potential side effects, other vaccinations, visits to general practitioner or on call doctor, and hospitalizations. Every survey period is 14 days, starting from day 0 (inclusion).

Blood samples for influenza antibody testing are collected from all participants at day 14 and 42. Samples for further immunological analyses are collected from subgroups at day 0, day 14, day 21, and day 42.

Vaccination schedule:

| Group | Day 0 (one shot) | Day 14 (two shots) | Day 42 |
|-------------|------------------|--------------------|-----------------|
| 1 | BCG | IIV + Placebo | Follow up visit |
| 2 (Control) | Placebo | IIV + Placebo | Follow up visit |
| 3 | Placebo | IIV + BCG | Follow up visit |
| 4 | IIV | Placebo + BCG | Follow up visit |

#### Randomization

Randomization takes place at baseline after informed consent is given. The randomization is done in varying blocks of 6-8, stratified by sex and age group (65-74; 75+) using REDCap



#### SAP BCG-DENMARK-ELDERLY, version 2.0, 08-06-2023



electronic data capture tools hosted at the Region of Southern Denmark<sup>[12,13]</sup>. As described above, participants are randomized to one of the four groups and given the allocated treatment.

#### Sample size

We aim to include 75 participants in each group, 300 in total. With an anticipated seroconversion rate of 50% in the control group, we should be able to show a 30% increase in seroconversion rate associated with BCG vaccine with 80% power and an alpha of 0.05, anticipating 10% loss to follow-up.

All participants are followed for clinical symptoms for six months. With this sample size, we will only be able to show differences in clinical symptoms if such differences are pronounced.

## Timing of final analyses and outcome assessments

All outcomes are analyzed after end of trial.

#### 11.0 STATISTICAL PRINCIPLES

## Levels of confidence and p-values

A double-sided p-value of < 0.05 will be considered statistically significant. 95% confidence intervals will be provided.

## **Protocol violations**

Protocol deviations and exclusions will be reported for each treatment arm.

#### 12.0 STUDY POPULATION

## **Screening data**

As described for part A.

### Recruitment

As described for part A.

## Exclusion/lost to follow-up



#### SAP BCG-DENMARK-ELDERLY, version 2.0, 08-06-2023



Participants who are excluded after randomization or lost to follow up are not replaced.

Participants are under follow-up for six months post-randomization or until they withdraw their consent, migrate to another country, or die.

## Baseline characteristics, study population

Continuous baseline characteristics will be reported as mean and standard deviation or median and inter-quartile range, as appropriate. Categorical baseline characteristics will be reported as count and percentage. No statistical testing for baseline characteristics will be performed.

#### 13.0 DESCRIPTION OF OUTCOMES AND VARIABLES

#### **Primary outcome**

Change in antibody levels to influenza virus strains included in the IIV, comparing levels at day 14 and day 42; just before and 4 weeks after influenza vaccination (for group 4, it will be 2 and 6 weeks after influenza vaccination).

We will use *Influvactetra* (Mylan ApS, Copenhagen), a quadrivalent inactivated influenza vaccine containing the following strains:

- 1. A/Victoria/2570/2019, IVR-215 (H1N1, pdm09-like strain)
- 2. A/Cambodia/e0826360/2020, IVR-224 (H3N2-strain)
- 3. B/Washington/02/2019, wild type
- 4. B/Phuket/3073/2013, wild type

Influenza antibodies are measured in hemagglutination-inhibition assay (HAI) $^{[22]}$  yielding dilution titers with an expected range of <20 to 320 for this population. Geometric mean titers (GMT) will be determined by calculating the mean of the log-transformed duplicate titers followed by back transformation (calculated as 10x, where x is defined as the mean log-transformed titer).

Seroconversion is defined as a pre-vaccination HAI titer <10 and a post-vaccination titer  $\geq$  40, or a pre-vaccination titer  $\geq$  10 and a minimum four-fold rise in post-vaccination titer<sup>[22]</sup>.

#### **Secondary outcomes**

Self-reported infections:





Infections are identified through information given by the participants in the electronic follow-up questionnaires, where they are asked to describe disease episodes every 14 days. They are asked if they have been ill, and then asked to cross of their symptoms on a list. Furthermore, we ask them to provide the most likely cause for their illness.

Disease episodes are characterized as infections if participants report symptoms compatible with an infectious disease or they report an infectious disease diagnose as the cause of their illness. Criteria for self-reported infection:

- Having one or more of the following symptoms: fever, cough, sore throat, runny nose/nasal congestion (common cold symptoms), loss of smell or taste sense, vomiting, or diarrhea with or without general symptoms such as headache, myalgia, dysarthria, or fatigue.
- Having dyspnea AND fever with or without general symptoms such as headache, myalgia, dysarthria, or fatigue.
- Having described an infectious disease as the self-estimated cause of illness. This is a
  free-text field and participants answers will be classified as infectious disease or not by
  medically trained study personnel.

Baseline for analysis is set at day 14 reflecting completion of the allocated vaccinations. We will however also conduct the analysis from day 0-14. Participants can register a maximum of one infectious disease event per survey period (14 days).

A secondary analysis of association between influenza antibody level and subsequent risk of infection will be performed to test if high antibody titers correlate with risk of infection.

*Immunological outcomes (subgroup analyses):* 

A random subset of participants (the first to accept) have extra blood samples taken for further immunological analyses.

- 1. Lymphocyte-dependent responses 7 days after influenza vaccination
- 2. The induction of innate immune memory 14- and 42-days post-randomization

For the lymphocyte analyses, 10 participants from groups 1-3 will have blood drawn on day 21, exactly 7 days after influenza vaccination. We will assess the effect of the different treatment combinations on the response to the influenza vaccine, examining activated





influenza antibody-secreting B-lymphocytes. Due to the different timing of the influenza vaccination, participants from group 4 are not part of this analysis.

For the trained immunity analyses, 15 participants from each group will have extra blood samples taken on day 0, 14, and 42. Peripheral blood mononuclear cells (PBMCs) are isolated from the samples and subsequently stimulated in vitro with various antigens. The immune function will be assessed by cytokine production capacity measured by Luminex technology after stimulation. The outcome measure for this analysis is concentration of different types of cytokines produced following stimulations. We will compare fold change in cytokine production between the groups at the various timepoints with and without adjustment for responses in control medium. This will allow us to determine whether BCG in the different combinations with influenza vaccine induces trained immunity in this population.

#### **List of variables:**

| Variable name | Definition | Туре | Scale |
|---|---|---|---|
| Primary outcome: Change in antibody levels to influenza virus strains included in the IIV, comparing levels at day 14 and day 42. | | | |
| ab_diff_strain | Influenza antibody titer (GMT) day 42 minus day 14. For each strain. | Continuous | <20 to 320 |
| seroconv | Seroconverted after influenza vaccination (4-fold increase in Ab titer). For each strain. | Binary | 0: no<br>1: yes |
| Secondary outcome | ome, self-reported infections: | - | 1 |
| infection | Infection or symptoms consistent with infection (0 or 1 every survey period). | Binary | 0: no<br>1: yes |
| Secondary expo | sure: | -1 | |
| ab_day42_cat | Influenza ab titer day 42 (GMT).<br>Secondary exposure. | Categorical | 1. quartile 2. quartile 3. quartile 4. quartile |
| Secondary outcome | ome, immunological: | | |
| b_lymph | Number of activated B-cells. For all relevant subtypes. | Continuous | 0.0-0.3 x<br>10 <sup>9</sup> /L |





| cytokine_stim | Cytokine concentration (TNF $\alpha$ , IL-1 $\beta$ , IFN- | Continuous | 0-1500 |
|---|---|---|---|
| _day | γ) after stimulation with: Poly(I:C), | | pg/mL |
| | Pam3CSK4, LPS, and influenza vaccine at | | |
| | the various timepoints (day 0, 14, and | | |
| | 42). | | |
| diff_cytokine_ | Fold change in cytokine concentration | Continuous | 0-10 |
| stim_day | from baseline value (day 0) to day 14 and | | |
| | 42 after stimulation with various stimuli. | | |
| | Compared between the randomization | | |
| | groups. Using randomization group as | | |
| | exposure (categorical). | | |

#### 14.0 ANALYSIS

#### Methods

All analyses will be performed from the intention-to-treat principle, for all participants studied together and stratified by sex and age group.

## **Primary outcome:**

Mean change in GMT in samples from day 14 and 42 will be compared between the control group and the three treatment groups in linear regression analyses with adjustment for baseline level of GMT, age group, and sex. In case residuals are not normally distributed, the analysis will be performed on log-10 transformed change in GMT instead. The proportion of participants who seroconvert will be compared in logistic regression analysis with adjustment for age group and sex.

## **Secondary outcomes:**

## *Self-reported infections:*

The hazard ratio of infections will be estimated using an Andersen-Gill Cox proportional hazards regression model with infections included as recurrent events and time since inclusion as underlying time scale. The proportional hazards assumption will be tested using Schoenfeld residuals. As participants are only able to report one infectious episode during a follow-up questionnaire, the event will be assigned to the first day within the questionnaire period, and the following 14 days of follow-up excluded for analyses as it represents risk free time.



#### SAP BCG-DENMARK-ELDERLY, version 2.0, 08-06-2023



Association between influenza antibody titer level at day 42 and rate of infections will also be explored in Andersen-Gill Cox proportional hazards regression model, using antibody titer at day 42 as exposure and self-reported infections after day 42 as outcome. Antibody titers will be categorized into quartiles or similar relevant categories. The analysis will be adjusted for sex and age group.

Absolute risk reduction will be calculated using Cox regression.

Immunological outcomes (subgroup analyses):

Mean change in number of activated B-cells, concentration of cytokines, as well as fold change in cytokine concentration after stimulation from day 0 to day 14 and from day 14 to day 42 will be compared between the control group and the three treatment groups in linear regression analyses. With and without adjustment for responses in the control condition.

## Missing data

Participants will be included in the analysis of the primary outcome irrespective of missing questionnaires as this is based on laboratory outcomes only. Participants with missing or inadequate blood samples on one of the sample days will be excluded from the antibody analysis.

For the secondary outcome (infection) which is based on self-reported information, participants are only under follow-up during the periods where they have completed follow-up questionnaires.

#### Adverse events

Adverse events will be described in terms of incidence in the randomization groups and more thoroughly presented in a table as part of supplementary material (Table 4). Serious adverse events (SAE) will be classified as related to study drugs (possible/probable/definite) or unrelated to study drugs (unlikely/doubtful). If related, they are classified as expected/unexpected (SAR/SUSAR).

#### 15.0 SUPPLEMENTARY INFORMATION

## Figures and tables

Figure 1: Flow chart, inclusion.







Figure 2: Study design.

Table 1: Baseline characteristics.

Table 2: Results primary outcome.

Table 3: Results infectious disease rate and association with influenza antibody level.

Figure 3: Results trained immunity.

Figure 4: Results lymphocyte response.

Table 4: Adverse events (AE) and Serious Adverse Events (SAE).

Table 5: Short description of Serious Adverse Events (SAE).





Figure 1: Flow chart, inclusion.







# Figure 2: Study design.

A flow chart describing enrollment, follow-up visits, vaccinations, collection of blood samples, and surveys with a timeline.





## Table 1: Baseline characteristics.

| | Group 1 | Group 2 | Group 3 | Group 4 |
|---|---|---|---|---|
| Age, median (IQR) | | | | |
| Sex female (%) | | | | |
| Living alone (%) | | | | |
| Spouse included in study (%) | | | | |
| Active smoker (%) | | | | |
| Previous smoker (%) | | | | |
| Alcohol consumption, units per week, mean (SD) | | | | |
| BMI, median (IQR) | | | | |
| Chronic diseases | | | | |
| Cardiovascular (%) | | | | |
| Diabetes (%) | | | | |
| Lung (%) | | | | |
| Other (%) | | | | |
| Level of education | | | | |
| Low (%) | | | | |
| Medium (%) | | | | |
| High (%) | | | | |
| Previously BCG vaccinated (%) | | | | |
| Scar from BCG vaccination observed (%) | | | | |
| COVID-19 vaccinated, yes (%) <sup>1</sup> | | | | |
| One dose | | | | |
| Two doses | | | | |
| Three doses | | | | |

<sup>&</sup>lt;sup>1</sup>COVID-19 vaccinated before enrollment.





# Table 2: Results primary outcome.

Change in antibody levels to influenza virus strains included in the IIV, comparing levels at day 14 and day 42.

| Influenza strain | Change in antibody titer from day 14 to day 42, mean (sd) $\beta \ (95\% \ \text{CI})$ | | | |
|---|---|---|---|---|
| | Group 1 | Group 2<br>(Control) | Group 3 | Group 4 |
| A/Victoria | xx (xx-xx) | xx (xx) | xx (xx) | xx (xx) |
| | xx (xx-xx) | (ref.) | xx (xx-xx) | xx (xx-xx) |
| A/Cambodia | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | xx (xx-xx) | (ref.) | xx (xx-xx) | xx (xx-xx) |
| B/Washington | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | xx (xx-xx) | (ref.) | xx (xx-xx) | xx (xx-xx) |
| B/Phuket | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | xx (xx-xx) | (ref.) | xx (xx-xx) | xx (xx-xx) |
| | | | ersion N (%)<br>95% CI) | |
| A/Victoria | xx (%) | xx (%) | xx (%) | xx (%) |
| | x.xx(x.xx–x.xx) | (ref.) | x.xx (x.xx–x.xx) | x.xx (x.xx–x.xx) |
| A/Cambodia | xx (%) | xx (%) | xx (%) | xx (%) |
| | x.xx(x.xx–x.xx) | (ref.) | x.xx (x.xx–x.xx) | x.xx (x.xx–x.xx) |
| B/Washington | xx (%) | xx (%) | xx (%) | xx (%) |
| | x.xx(x.xx–x.xx) | (ref.) | x.xx (x.xx–x.xx) | x.xx (x.xx–x.xx) |
| B/Phuket | xx (%) | xx (%) | xx (%) | xx (%) |
| | x.xx(x.xx-x.xx) | (ref.) | x.xx (x.xx–x.xx) | x.xx (x.xx–x.xx) |



Table 3: Results infectious disease rate and association with influenza antibody level.

| Treatment group | ment group Number Hazard (%) (95% | | Absolute risk<br>reduction<br>(95% CI) |
|---|---|---|---|
| Self-reported infection six months post-randomization | | | |
| Group 1 | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Group 2 | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Group 3 | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Group 4 | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| Association betwee | n influenza antibo | dy level at day 42 and in | fection rate during |
| | follow-up | after day 42 | |
| Antibody level by | Number | Hazard ratio | Absolute risk |
| quartile | (%) | (95% CI) | reduction<br>(95% CI) |
| 1 quartile | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| 2 quartile | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| 3 quartile | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |
| 4 quartile | xx (x.x) | x.xx (x.xx–x.xx) | x.x% (x.x%–x.x%) |



## Figure 3: Results trained immunity.

Boxplots showing fold increase in cytokine production after stimulation with bacterial antigens and influenza vaccine at day 0, day 14, and day 42 for each treatment group.



<sup>\*</sup> Denotes within-group statistically significant change in cytokine levels between day 0 and 14 or between day 14 and 42



Δ Denotes between group statistically significant different change in cytokine levels between day 0 and 14 or between day 14 and 42



# Figure 4: Results lymphocyte response.

Graphs showing numbers and or percentage of activated B-lymphocytes at day 21 per treatment group.





# Table 4: Adverse events (AE) and Serious Adverse Events (SAE).

| Endpoint | Treatment group | | | |
|---|---|---|---|---|
| | 1 | 2 | 3 | 4 |
| | Number (%)<br>[M/F] | | | |
| Any SAE | | | | |
| Hospitalization for any reason | | | | |
| Death due to any reason | | | | |
| Injection site reaction | | | | |
| Minor abscess/wound | | | | |
| Severe local reaction (abscess) | | | | |
| Fever | | | | |
| Fatigue | | | | |
| Headache | | | | |
| Lymphadenitis | | | | |
| Blood or lymphatic disorder | | | | |
| Cardiac disorders | | | | |
| Endocrine disorders | | | | |
| Gastrointestinal disorders | | | | |
| Infection | | | | |
| Musculoskeletal and connective tissue disorders | | | | |
| Nervous system disorders | | | | |
| Respiratory disorders | | | | |
| Urological and gynecological disorders | | | | |





## SAP BCG-DENMARK-ELDERLY, version 2.0, 08-06-2023

| Unknown/other |
|------------------------------------|
| Life threatening |
| Required/prolonged hospitalization |
| Resulted in death |



# **Table 5 Short description of Serious Adverse Events (SAE)**

| No | Category | Outcome | Description | Group <sup>1</sup> | Sex | Week <sup>2</sup> | Before/after <sup>3</sup> |
|---|---|---|---|---|---|---|---|
| 1 | | | | | | | |
| 2 | | | | | | | |
| 3 | | | | | | | |
| 4 | | | | | | | |
| 5 | | | | | | | |
| 6 | | | | | | | |
| 7 | | | | | | | |
| 8 | | | | | | | |
| 9 | | | | | | | |
| 10 | | | | | | | |

<sup>&</sup>lt;sup>1</sup>Randomisation group.

<sup>&</sup>lt;sup>2</sup>Weeks after inclusion.

<sup>&</sup>lt;sup>3</sup>Occurrence before or after other vaccines were administered to the participant.



#### **16.0 REFERENCES**

- 1. United Nations, Department of Economic and Social Affairs, Population, Division . World Population Ageing 2015. 2015;(ST/ESA/SERA/390).
- 2. Crooke SN, Ovsyannikova IG, Poland GA, Kennedy RB. Immunosenescence and human vaccine immune responses. Immun Ageing 2019;16(1).
- Higgins JPT, Soares-Weiser K, López-López JA, Kakourou A, Chaplin K, Christensen H, et al. Association of BCG, DTP, and measles containing vaccines with childhood mortality: Systematic review. BMJ 2016;355.
- 4. Kristensen I, Aaby P, Jensen H, Fine P. Routine vaccinations and child survival: follow up study in Guinea-Bissau, West Africa Commentary: an unexpected finding that needs confirmation or rejection. BMJ 2000;321(7274):1435–1435.
- 5. Benn CS, Fisker AB, Rieckmann A, Sørup S, Aaby P. Vaccinology: time to change the paradigm? Lancet Infect Dis 2020;20(10):e274–83.
- 6. Netea MG, Quintin J, Van Der Meer JWM. Trained immunity: A memory for innate host defense. Cell Host Microbe 2011;9(5):355–61.
- 7. Netea MG, Joosten LAB, Latz E, Mills KHG, Natoli G, Stunnenberg HG, et al. Trained immunity: A program of innate immune memory in health and disease. Science (80-.).2016;352(6284):427.
- [Kleinnijenhuis J, Quintin J, Preijers F, Joosten LAB, Ifrim DC, Saeed S, et al. Bacille Calmette-Guérin induces NOD2-dependent nonspecific protection from reinfection via epigenetic reprogramming of monocytes. Proc Natl Acad Sci U S A 2012;109(43):17537– 42.
- Giamarellos-Bourboulis EJ, Tsilika M, Moorlag S, Antonakos N, Kotsaki A, Domínguez-Andrés J, et al. Activate: Randomized Clinical Trial of BCG Vaccination against Infection in the Elderly. Cell 2020;183(2):315-323.e9.
- 10. Tsilika M, Taks E, Dolianitis K, Kotsaki A, Leventogiannis K, Damoulari C, et al. ACTIVATE-2: A Double-Blind Randomized Trial of BCG Vaccination Against COVID-19 in Individuals at Risk. Front Immunol 2022;13:873067.
- 11. O'Neill LAJ, Netea MG. BCG-induced trained immunity: can it offer protection against COVID-19? Nat Rev Immunol 2020;20(6):335–7.





- 12. Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, et al. The REDCap consortium: Building an international community of software platform partners. J. Biomed. Inform.2019;95.
- 13. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)-A metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform 2009;42(2):377–81.
- 14. Dorrington MG, Bowdish DME. Immunosenescence and novel vaccination strategies for the elderly. Front. Immunol.2013;4(JUN).
- 15. Goodwin K, Viboud C, Simonsen L. Antibody response to influenza vaccination in the elderly: A quantitative review. Vaccine 2006;24(8):1159–69.
- Chen WH, Kozlovsky BF, Effros RB, Grubeck-Loebenstein B, Edelman R, Sztein MB.
   Vaccination in the elderly: an immunological perspective. Trends
   Immunol.2009;30(7):351–9.
- 17. Biering-Sørensen S, Aaby P, Lund N, Monteiro I, Jensen KJ, Eriksen HB, et al. Early BCG-Denmark and Neonatal Mortality among Infants Weighing <2500 g: A Randomized Controlled Trial. Clin Infect Dis 2017;65(7):1183–90.
- 18. Cirovic B, de Bree LCJ, Groh L, Blok BA, Chan J, van der Velden WJFM, et al. BCG Vaccination in Humans Elicits Trained Immunity via the Hematopoietic Progenitor Compartment. Cell Host Microbe 2020;
- 19. Libraty DH, Zhang L, Woda M, Acosta LP, Obcena A, Brion JD, et al. Neonatal BCG vaccination is associated with enhanced T-helper 1 immune responses to heterologous infant vaccines. Trials Vaccinol 2014;3(1):1–5.
- 20. Ritz N, Mui M, Balloch A, Curtis N. Non-specific effect of Bacille Calmette-Guérin vaccine on the immune response to routine immunisations. Vaccine 2013;31(30):3098–103.
- 21. Leentjens J, Kox M, Stokman R, Gerretsen J, Diavatopoulos DA, Van Crevel R, et al. BCG vaccination enhances the immunogenicity of subsequent influenza vaccination in healthy volunteers: A randomized, placebo-controlled pilot study. J Infect Dis 2015;212(12):1930–8.
- 22. Katz JM, Hancock K, Xu X. Serologic assays for influenza surveillance, diagnosis and vaccine evaluation. Expert Rev. Anti. Infect. Ther.2011;9(6):669–83.

